CLINICAL TRIAL: NCT05032716
Title: Treadmill Training is an Effective Rehabilitation Program in Treatment of Children With Acute Lymphoblastic Leukemia
Brief Title: EFFECT OF TREADMILL TRAINING ON BALANCE AFTER CHEMOTHERAPY IN CHILDREN WITH ACUTE LYMPHOBLASTIC LEUKEMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/ 012/001956
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance exersices group (Active Comparator): received traditional exercise program with instructions given to the children for 60 min aiming to improve posture control and balance
  Interventions: Other: Balance exrcises
- Balance exersices and treadmill group (Active Comparator): received the same traditional physical therapy program as the same applied in group of balance exercise (30 min), in addition to treadmill training (30 min)
  Interventions: Other: Balance exrcises and Treadmill training

INTERVENTIONS:
Other: Balance exrcises — the group (20 children) received traditional exercise program with instructions given to the children for 60 min aiming to improve posture control and balance. Tools of traditional physical therapy exercises were; special tools were used for traditional physical therapy exercises include vestibular board, rolls of different sizes, blocks and wedges of different heights
  Arms: Balance exersices group
Other: Balance exrcises and Treadmill training — the group (20 children) received the same traditional physical therapy program as the same applied in group of balance exercises, in addition to treadmill training (30 min). The child walked on the treadmill (motorized treadmill, ENTRED, Enraf-Nonius) at 75% of over-ground speed and individually prescribed low-endurance walking at 0% incline for 20 min, three times a week for 8 successive weeks. The walking area of the treadmill is made from heavy steel with a minimum 8-inch thickness and is available with cushioning in case of accidental impacts. Before the walking session, each child underwent 5 min of active stretching exercises that include prolonged and progressive stretching of the hamstrings, quadriceps muscles, and Achilles tendon.
  Arms: Balance exersices and treadmill group

SUMMARY:
Purpose: The present research was conducted to study the effect of treadmill training on balance after chemotherapy in children with acute lymphoblastic leukemia.

Subjects and Methods: Forty children with acute lymphoblastic leukemia included in the current research ranged of age from 8 to 12 years. The children participated in this study were assigned randomly into two equal number groups (A and B). Group (A) includes 20 children who received balance exercises, while group (B) includes 20 children who received the same balance exercises of group (A) and treadmill training. The treatment program was applied three sessions per week (60 min for every session) for 8 weeks. Balance Master System and Biodex Balance System were used to evaluate balance of all children in the three groups before and after the treatment program.

DETAILED DESCRIPTION:
The current research is a randomized control trial to differentiate between the treadmill training on balance after chemotherapy in children with acute lymphoblastic leukemia. Chemotherapy induced peripheral neuropathy is related to the intensity of treatment and dosage of chemotherapy which could affect the severity of its symptoms, it could result in serious problems like sensory changes and numbness , in case the sensory nerves were affected , muscle weakness and in-coordination in case the affected were the motor nerves. In addition to the psychological problems the patient experience as a result of CIPN, the patient also experience physical problems like injuries, fear of fall results from lack of sensory perception and muscle power. Treadmill training, motor training may favor proprioceptive feedback, leading to adjustments for adequate postural balance and functional performance. Treadmill exercises stimulate the kinetic, kinematic, and temporal features of walking. These exercises improve the strength of the muscles of the lower extremities, enhance motor learning, improve functional abilities, and activate the locomotor control system

ELIGIBILITY:
Inclusion Criteria:

* able to recognize commands given to them,
* understand our verbal command and encouragement,
* and stand and walk independently without repeated falling

Exclusion Criteria:

* Children with impairment of sensation or
* other neurological or psychological problems,
* tightness and/or fixed deformity of lower limbs,
* any neurological, musculoskeletal, or mobility disorders,
* cardiac anomalies,
* vision or hearing loss

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
Step/Quick Turn (SQT) | 2 months
  Turn Time (sec) from right and left side
Step/Quick Turn | 2 months
  Turn Sway (deg/sec) from right and left side
Tandem Walk (TW) | 2 months
  to measure Speed (cm/sec)
Tandem Walk (TW) | 2 months
  to measure End Sway (deg/sec)
Overall Stability Index | 2 months
  from Biodex Balance System
Antero-posterior Stability Index | 2 months
  from Biodex Balance System
Medio-lateral Stability Index | 2 months
  from Biodex Balance System

CONTACTS AND LOCATIONS:
Overall Officials: Reham Alsakhawi, Ph.D, Principal Investigator — Assistant Professor, Faculty of Physical Therapy, Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate
  - Faculty of Physical Therapy, Giza

IPD SHARING:
Plan to Share IPD: Yes
data from participants will be made available
Supporting Information: Study Protocol
Time Frame: 6 months after study completion
Access Criteria: data access requests will be reviewed by an external independent review panel. requestor will be required to sign a data access agreement